CLINICAL TRIAL: NCT01645943
Title: Randomized Comparison Between Invasive and Conservative Strategies in Patients With Non-ST-segment Elevation Acute Coronary Syndrome and Comorbidities
Brief Title: Invasive vs Conservative Strategies in Non-ST-elevation Acute Coronary Syndrome and Comorbidities
Acronym: MOSCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Juan Sanchis, Full Professor of Medicine, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/ 01595
Record Dates: First submitted 2012-07-13; First posted 2012-07-20 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Acute Coronary Syndrome
Keywords: Non-ST-elevation acute myocardial infarction; Comorbidities
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conservative (No Intervention): Coronary angiogram only if recurrent ischemia or peristent heart failure or inducible ischemia in predischarge stress test if perfomed
- Invasive (Active Comparator): Routine coronary angiogram
  Interventions: Procedure: Coronary angiogram

INTERVENTIONS:
Procedure: Coronary angiogram — Routine coronary angiogram and revascularization if indicated
  Arms: Invasive

SUMMARY:
The guidelines of clinical practice, based on the randomized studies, recommend an invasive strategy in non-ST elevation acute coronary syndrome (NSTEACS). However, patients with comorbidities are excluded from the randomized studies and the observational registries showthat patients with comoribidities undergo fewer cardiac catheterizations. The aim is to investigate the benefit of the invasive strategy in patients with NSTEACS and comorbidities.

Patients hospitalized with NSTEACS, older than 70 years and with significant comorbidities, will be included. The latter will be defined as at least 2 of the following: peripheral artery disease, cerebral vascular disease, dementia, chronic pulmonary disease, chronic renal failure and anemia. The included patients will be randomized to an invasive (routine coronary angiogram) or conservative (coronary angiogram only if recurrent or inducible ischemia) strategy. All patients will receive medical treatment according to current recommendations.

The main outcome will be death, reinfarction or readmissions by heart cause at one-year follow-up. The hypothesis is that an invasive strategy will improve prognosis in patients with NSTEACS and comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Age =>70 years old
* Angina chest pain
* Troponin elevation
* At least 2 of the following comorbidities: A) Documented peripheral artery disease. B)Renal filaure (GFR <45 ml/min/m2). C) Neurological disease with permanent deficit. D) Dementia (Pfeiffer test). E) Chronic pulmonary disease (Gold>2 or ambulatory oxigen therapy). Anemia (Hb =<11 g/dl)

Exclusion Criteria:

* Dynamic ST changes (=>1 mm) in the initial ECG
* Prior known non-revascularizable coronay disease
* Concomitant heart disease different to coronary disease
* Life expentancy < 1 year

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 109 (Actual)
Dates: Start 2012-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
All cause mortality, reinfarction or reasmission by cardiac cause | 1 year

SECONDARY OUTCOMES:
Days alive out of the hospital | 1 year
Bleeding | In-hospital (average= 1 week)
Renal failure | In-hospital (average= 1 week)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Sanchis, Full Prof, Principal Investigator — University of Valencia. University Clinic Hospital
Locations (6):
- Spain (6):
  - Hospital Pujol i Trias, Badalona, Barcelona
  - Hopsital Clinic, Barcelona, Barcelona
  - Hospital Virgen del Rosell, Cartagena, Murcia
  - Hospital Clínico Universitario, Valencia, Valencia
  - Hospital Valle Hebrón, Barcelona
  - Hospital Virgen Arrixaca, Murcia

REFERENCES:
- [Result] Sanchis J, Nunez E, Barrabes JA, Marin F, Consuegra-Sanchez L, Ventura S, Valero E, Roque M, Bayes-Genis A, Del Blanco BG, Degano I, Nunez J. Randomized comparison between the invasive and conservative strategies in comorbid elderly patients with non-ST elevation myocardial infarction. Eur J Intern Med. 2016 Nov;35:89-94. doi: 10.1016/j.ejim.2016.07.003. Epub 2016 Aug 8. PMID 27423981